CLINICAL TRIAL: NCT04714853
Title: Pilot Study to Determine the Effect of Different Dialysis Treatment Modalities and Diet on Gastrointestinal Bacteria and Azotaemic Toxins
Brief Title: Different Dialysis Modalities and Diet on Gastrointestinal Biome and Azotaemic Toxins
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University of Brighton (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0308
Record Dates: First submitted 2016-02-10; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Kidney Failure
Keywords: microbiome; haemodialysis; peritoneal dialysis
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
. This is a prospective observational pilot study to analyse gastrointestinal tract bacterial populations in peritoneal dialysis and haemodialysis patients under the care of the Royal Free Hospital with chronic kidney disease who have been established on regular haemodialysis and peritoneal dialysis treatments in a Royal Free Hospital kidney care centre.

DETAILED DESCRIPTION:
Patients, attending for outpatient haemodialysis and peritoneal dialysis to be tested for gastrointestinal tract bacterial population by taking a single mouth swab, and a stool sample. Additional blood sampling, when patients are having blood tests for routine clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years and older up to 80 years
* Under the care of the Royal Free Hospital with chronic kidney disease and established on regular haemodialysis or peritoneal dialysis.
* Able to provide written informed consent obtained

Exclusion Criteria:

* Patients unable to provide written informed consent
* Patients not fulfilling inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 dialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2023-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
generation of bacterial phylogenetic trees by identifying different bacteria from stool samples and oral swabs by analysis of bacterial ribosomal 16S | 5 years
  observational

SECONDARY OUTCOMES:
measure indoxyl sulphate (IS) and p-Cresyl sulfate (PCS) umol/L | 8 years
  observational

CONTACTS AND LOCATIONS:
Overall Officials: andrew davenport, Principal Investigator — UCL Centre for Nephrology, Royal Free Hospital
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
data to be deposited with UCL